CLINICAL TRIAL: NCT04755036
Title: National Survey and Case-vignette Study of Clinical Decisions in Pancreatic Cancer
Acronym: GECP01
Status: Completed | Type: Observational
Sponsor: Hospital Miguel Servet (Other)
Collaborators: Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, Mario Serradilla, MD, FACS, Senior Consultant in Department of Surgery, Hospital Miguel Servet
Other Study IDs: HGUA01
Record Dates: First submitted 2021-01-15; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey and case vignette — We sent a survey and case vignette cases to every responsible in each center

SUMMARY:
Very few surveys have been carried out about oncosurgical decisions made in patients with pancreatic cancer (PC), and none have established whether the therapeutic approaches differ between low/medium and high volume centers.

A survey was sent out to centers from Spanish Group of Pancreatic Surgery (GECP) asking about usual pre, intra and postoperative management of PC patients and describing five imaginary cases of PC corresponding to common scenarios that surgeons regularly assess in oncosurgical meetings. Investigators define consensus when 80% of answers were equal.

DETAILED DESCRIPTION:
In 2019, the Hepato-Pancreato-Biliary Surgery Section of the Spanish Association of Surgeons and the Spanish Chapter of the IHPBA created the Spanish Group of Pancreatic Surgery (henceforth, GECP). The GECP notified the associates of both societies about the creation of the group by email, and also made announcements on their respective web pages. The GECP comprises a council of eight people. On applying to join, hospitals appoint a contact person who receives information on the work of the group, which is carried out on a multicenter basis. Currently, 72 hospitals are part of the GECP. GECP members perform 78% of PDs throughout Spain.

In January 2020, a survey was sent out to the local surgeon manager of each GECP center, describing decisions in pre, intra, and postoperative management of patients with PC undergoing PD and five imaginary cases of patients with PC in the pancreatic head corresponding to five common scenarios that surgeons regularly assess in multidisciplinary oncological meetings (MDTB). It was explained in the cover letter that respondents' answers should not necessarily be the ones that appear in the textbooks or clinical guidelines but should reflect standard clinical practices at their centers. In the interests of objectivity, it was decided that the responses should be anonymous. The questions about decisions and cases were devised by the first author and sent to the seven other members of the GECP organizing committee who evaluated them and finally agreed on their definitive format. The cases presented were: resectable PC without vascular invasion, resectable PC with venous invasion below 180º, borderline PC with venous invasion above 180º, PC with arterial invasion below 180º and severe venous invasion, and PC with liver metastases.

Investigators classified hospital level divided as follows (level 1: 0-250 beds or area <200,000 inhabitants; level 2: 251-500 beds or area <400,000; level 3: > 500 beds or area> 400,000); whether liver transplantation is performed at the center (to assess whether greater experience in vascular reconstruction affected intraoperative vascular management); the number of hospital beds; the number of pancreaticoduodenectomies (PD), distal pancreatectomies (DP) and total pancreatectomies (TP) performed at each center in 2018; and data on the surgeon who completed the survey including age, gender, position and years of experience in pancreatic surgery. Respondents were given a period of 60 days to submit their replies.

The data were collected through an electronic survey using Google Forms and were analyzed with the R statistical software (https://www.r-project.org/). Categorical variables were expressed as number of cases and percentages. For continuous variables, normality was assessed with the Shapiro-Wilk test. Variables that were normal were expressed by means and standard deviation, while those that deviated from normality were expressed with medians and interquartile range. As contrast tests, the chi-square test with Yates correction was used for categorical variables, and the Student's t test and the Mann-Whitney U test for continuous normal and non-normal variables respectively. We defined the existence of a common national criterion when 80% of the respondents applied the same clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Resposnible for each center of GECP

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surgeons responsible of GECP in each center
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of consensus in therapeutical decisions in pancreatic cancer between low/mid vs high volume hospitals | Survey sent in 2020. Time to receive surveys up to 12 weeks
  Percentage of consensus in therapeutical decisions. Difference (p<0.05) (if exists) between high and low volume centers

CONTACTS AND LOCATIONS:
Overall Officials: Jose Ramia, PhD, Principal Investigator — Hospital General Universitario de Alicante
Locations (1):
- Jose M Ramia, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramia JM, Cugat E, De la Plaza R, Gomez-Bravo MA, Martin E, Munoz-Bellvis L, Padillo FJ, Sabater L, Serradilla-Martin M. Clinical decisions in pancreatic cancer surgery: a national survey and case-vignette study. Updates Surg. 2023 Jan;75(1):115-131. doi: 10.1007/s13304-022-01415-1. Epub 2022 Nov 14. PMID 36376560